CLINICAL TRIAL: NCT06103097
Title: "Assessment of the Histological Evolution of Pediatric Patients With Liver Transplantation"
Brief Title: Histologic Evolution of Patients With Liver Transplantation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Vall d'Hebron (Other)
Collaborators: Sociedad Espanola de Gastroenterologia, Hepatologia y Nutricion Pediatrica (Other)
Responsible Party: Principal Investigator, Jesús Quintero, Lead Clinician; Pediatric Hepatology and Liver Transplant Department, Hospital Vall d'Hebron
Other Study IDs: PR(AMI)511/2018
Record Dates: First submitted 2023-10-15; First posted 2023-10-26 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Liver Transplant Failure and Rejection; Children, Only
Keywords: Liver Histology; Follow-up Liver Biopsy
MeSH Terms: conditions — Rejection, Psychology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chohort of pediatric Liver transplant pacients: Patients under 18 years recipient of a Liver transplanbt followed in our Unit and under the follow-up liver biopsy protocol
  Interventions: Other: No interventions done (obervational)

INTERVENTIONS:
Other: No interventions done (obervational) — Observational study

SUMMARY:
Certain pediatric liver transplant patients with immunosuppression levels in the therapeutic range and normal liver function tests present histological alterations (inflammation or fibrosis) in protocol biopsies.

The objective of the study was to evaluate the histological findings of protocol biopsies performed at 2, 5, 10 and 15 years after liver transplantation in pediatric patients. A follow-up biopsy is also performed 1 and 3 years after liver rejection.

To do that, a cohort study will be carried out by collecting clinical, analytical and histological data of patients undergoing post-liver transplant follow-up in pediatric hepatology and liver transplant outpatient clinics. According to the follow-up protocol for these patients, a liver biopsy is performed at 2, 5, 10 and 15 years after the transplant. In addition, ultrasound, elastography and general analysis with autoimmunity and HLA studies are carried out.

The evaluation of the histological evolution of the liver graft and its relationship with clinical and analytical changes will favor the management of immunosuppressive treatment in pediatric patients with liver transplants.

DETAILED DESCRIPTION:
Given the increase in survival of both the graft and the transplanted patient, new questions arise regarding long-term follow-up. In general, transplant patients undergo follow-up visits that include blood tests and abdominal ultrasounds. Immunosuppression levels, graft function and possible complications (infectious, tumorous, acute or chronic rejection, renal) are monitored.

The use of immunosuppressants is mainly associated with renal, infectious complications and de novo cancer. However, insufficient levels of immunosuppression can lead to graft rejection. On the one hand, various authors have attempted to completely withdraw immunosuppressive treatment in selected patients. On the other hand, histological alterations have been evidenced in patients with normal liver function tests and who maintained serum levels of immunosuppression in the therapeutic range. The balance between these two situations in not always easy.

Hypothesis:

Certain pediatric liver transplant patients with immunosuppression levels in the therapeutic range and normal liver function tests present histological alterations (inflammation or fibrosis) in protocol biopsies.

Main objetive:

To evaluate the histological findings of protocol biopsies performed at 2, 5, 10 and 15 years after liver transplantation in pediatric patients.

STUDY PROTOCOL:

Retrospective data collection through review of medical records of pediatric liver transplant patients who meet the inclusion criteria. For the protection of personal data, the data collection form will under no circumstances contain the name or NHC, only the date of birth, weight and gender of the patient will be referenced. Each patient will be uniquely identified by an identification number (ID) that will be automatically administered by the same computer program. The correlation between the coding and the patients' personal information will be kept in written format and under lock and key in the Vall d'Hebron Hospital facilities. The demographic, clinical, analytical, ultrasound, elastographic and biopsy data of the patients will be collected. With the data collected, a database will be created that allows its analysis. The platform used to collect said data will be Certain-Li, complying with the coding requirements for patient anonymity. This is a platform developed within the framework of the international working group Graft Injury Group observing long term outcomes.

LT Follow-Up All patients received immunosuppressant treatment according to our standard protocol in accordance with current European guidelines. To monitor graft function, liver function tests were measured every 2-3 months and Doppler Ultrasound was performed annually. Liver stiffness was assessed by transient elastography (TE) using FibroScan ® (Echosens, Paris, France) with a pediatric (S) or adult (M) probe, as appropriate. TE evaluations were performed annually and whenever a follow-up biopsy was performed.

Follow-up liver biopsies Follow-up liver biopsies were obtained from patients with normal liver function tests to control histopathological changes at 2, 5, 10, and 15 years after transplantation and just before transition to adult care (aged 18 to 20 years) Diagnosis of acute liver rejection was always made by biopsy (BPAR), and rejection was graded using the Rejection Activity Index (RAI) score according to the Banff classification The fibrosis stage was assessed using the ISHAK score (0-6) in every liver biopsy

Statistical study All data collected in this registry will be provided in patient data listings. Summary tables and/or graphs will be presented for the selected parameters as appropriate to the data.

For descriptive analyses, continuous patient variables will be expressed as mean and standard deviation or median and interquartile range depending on the nature of each variable. For continuous variables, the Sudent t test for independent samples will be used, or the Mann Whitney U test when the variable does not follow a normal distribution. Fisher's exact test or the Chi-square test was used for discrete variables. The differences will be considered statistically significant with a p<0.05 (two-sided contrast). To evaluate the correlation between the follow-up time and the different variables that show liver involvement, the Pearson or Spearman coefficient will be used depending on whether or not they follow a normal distribution, respectively. The correlation coefficients will be interpreted according to the guidelines of Fleiss et al, being classified as excellent when R > 0.75, good if 0.40 ≤ R ≤ 0.75, or poor if R < 0.40. Statistical analyzes will be performed using SPSS statistical software, version 18.0 (SPSS Corporation, Chicago, IL, USA).

ELIGIBILITY:
Inclusion Criteria:

* Patients between 2-18 years old who have received a liver transplant at least two years ago
* Follow-up in pediatric hepatology and liver transplant outpatient clinics at the Vall d'Hebron Hospital
* Performing tests, ultrasound, elastography and biopsy during the last year as part of the follow-up protocol of our center
* Patients who have signed the informed consent for inclusion in the study and the corresponding assents.

Exclusion Criteria:

* Patients who do not meet all the inclusion criteria of the protocol.
* Patients who are transplant recipients of multiple solid organs.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: - Patients under 18 years of age who have received an isolated liver transplant and who are currently being monitored in the Pediatric Liver Transplant Unit of the Vall d'Hebron University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-03-15 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Sublcinical inflamation | From 15 March 2019 to 31 december 2024
  Patients with normal liver function tests and RAI > 2 in the follow-up liver biopsy

SECONDARY OUTCOMES:
Fibrosis | From 15 March 2019 to 31 december 2024
  Any degree of fibrosis assessed using the ISHAK score observed in the follow-up liver biopsy
Sublcinical inflamation modification | From 15 March 2020 to 31 december 2024
  Change in the degree of inflamation (RAI) observed between the first follow-up liver biopsy and the 1 year control (in patients with biopsy proven actute rejection)

CONTACTS AND LOCATIONS:
Overall Officials: Jesus Quintero, MD, Principal Investigator — Responsible of Pediatric Hepatology and Liver Transplant Department
Locations (1):
- Hospital Universitari Vall d'Hebron, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No
IPD will be no available to other researchers

REFERENCES:
- [Result] Muiesan P, Vergani D, Mieli-Vergani G. Liver transplantation in children. J Hepatol. 2007 Feb;46(2):340-8. doi: 10.1016/j.jhep.2006.11.006. Epub 2006 Dec 1. PMID 17161491
- [Result] Feng S. Long-term management of immunosuppression after pediatric liver transplantation: is minimization or withdrawal desirable or possible or both? Curr Opin Organ Transplant. 2008 Oct;13(5):506-12. doi: 10.1097/MOT.0b013e328310b0f7. PMID 19060534
- [Result] Feng S, Ekong UD, Lobritto SJ, Demetris AJ, Roberts JP, Rosenthal P, Alonso EM, Philogene MC, Ikle D, Poole KM, Bridges ND, Turka LA, Tchao NK. Complete immunosuppression withdrawal and subsequent allograft function among pediatric recipients of parental living donor liver transplants. JAMA. 2012 Jan 18;307(3):283-93. doi: 10.1001/jama.2011.2014. PMID 22253395
- [Result] Feng S, Demetris AJ, Spain KM, Kanaparthi S, Burrell BE, Ekong UD, Alonso EM, Rosenthal P, Turka LA, Ikle D, Tchao NK. Five-year histological and serological follow-up of operationally tolerant pediatric liver transplant recipients enrolled in WISP-R. Hepatology. 2017 Feb;65(2):647-660. doi: 10.1002/hep.28681. Epub 2016 Jul 27. PMID 27302659